CLINICAL TRIAL: NCT03342742
Title: Daily Caloric Restriction and Intermittent Fasting in Overweight and Obese Adults With Autosomal Dominant Polycystic Kidney Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 17-1327; R03DK118215 (NIH)
Record Dates: First submitted 2017-10-27; First posted 2017-11-17 (Actual); Results first posted 2022-03-03 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-02

CONDITIONS: Polycystic Kidney, Autosomal Dominant
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Daily Caloric Restriction (Experimental): The daily caloric restriction group will be instructed to reduce energy intake by a 34% daily energy deficit from baseline individual weight maintenance energy requirements.
  Interventions: Behavioral: Weight Loss
- Intermittent Fasting (Experimental): Participants in the intermittent fasting group will be instructed to reduce energy intake to ~20% of estimated energy requirement (delivered as a single meal) three non-consecutive days per week, resulting in a weekly energy deficit of ~34% (similar to the daily caloric restriction group).
  Interventions: Behavioral: Weight Loss

INTERVENTIONS:
Behavioral: Weight Loss — Weight loss behavioral intervention via one of two strategies.

SUMMARY:
The proposed research will determine the feasibility of delivering two behavioral weight loss interventions for 1 year in adults with autosomal dominant polycystic kidney disease (ADPKD) who are overweight or obese. The study will also compare these two interventions in terms of safety, acceptability, and tolerability. Last, this pilot trial will provide initial insight into a) biological changes and b) changes in kidney growth with each of the two weight loss interventions.

DETAILED DESCRIPTION:
Autosomal dominant polycystic kidney disease (ADPKD) is characterized by development and continued growth of numerous fluid-filled renal cysts that ultimately result in renal failure. Similar to the general population, the prevalence of overweight and obesity have been rising in ADPKD patients, effecting about two-thirds of individuals. Surprisingly, the role of obesity in ADPKD progression is currently unknown. The investigators have novel preliminary data that overweight and obesity are independently associated with substantially faster kidney growth in ADPKD patients. Furthermore, in rodent models of ADPKD, mild-to-moderate food restriction profoundly slows cyst growth and maintains renal function via mechanisms including AMPK-activated kinase pathway activation and suppression of mammalian target of rapamycin/S6 kinase signaling and insulin-like growth factor-1 levels. Collectively, these data suggest that dietary restriction regimens may slow ADPKD progression. Accordingly, the primary aim is to determine the feasibility of delivering a 1 year behavioral weight loss intervention program in 30 overweight/obese adults with ADPKD, based on either daily caloric restriction (DCR) or intermittent fasting (IMF), with a similar (~34%) targeted weekly energy deficit. A key secondary goal is to evaluate safety, acceptability, and tolerability of IMF in ADPKD versus DCR. Last, the third exploratory aim is to a) obtain mechanistic insight into biological pathways that may be altered and b) provide initial insight into any changes in total kidney volume by magnetic resonance imaging with IMF and/or DCR.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-65 years
2. ADPKD diagnosis based on the modified Pei-Ravine criteria
3. BMI 25-45 kg/m^2
4. Normal to mildly declined renal function with an estimated glomerular filtration rate (eGFR) ≥30 mL/min/1.73 by the CKD-EPI equation
5. Access to the internet with video chat capabilities
6. No plans for extended travel (>2 weeks) during the 3 month intesive period
7. Not currently participating in another interventional study or weight loss program
8. Ability to provide informed consent

Exclusion Criteria:

1. Diabetes mellitus (diagnosis or fasting glucose >126 mg/dL or Hemoglobin A1C >6.5%)
2. Current nicotine use or history of use in the past 12 months
3. Alcohol or substance abuse (self-report or undergoing treatment)
4. History of hospitalization or major surgery within the last 3 months
5. Untreated dyslipidemia (low density lipoprotein cholesterol > 190 mg/dL or triglycerides >400 mg/dL)
6. Uncontrolled hypertension (systolic blood pressure > 160 or diastolic blood pressure >100 mm Hg)
7. Pregnancy, lactation, or unwillingness to use adequate birth control
8. Cardiovascular disease, peripheral vascular disease, cerebrovascular disease, significant pulmonary or gastrointestinal disease (described below), cancer (within the last 5 years, except skin cancer or other cancers considered cured with excellent prognosis)
9. Abnormal resting electrocardiogram (ECG): serious arrhythmias, including multifocal PVC's, frequent PVC's (defined as 10 or more per min), ventricular tachycardia (defined as runs of 3 or more successive PVC's), or sustained atrial tachyarrhythmia; 2nd or 3rd degree A-V block, QTc interval > 480 msec or other significant conduction defects
10. Significant gastrointestinal disorders including: chronic malabsorptive conditions, peptic ulcer disease, Crohn's disease, ulcerative colitis, chronic diarrhea, or active gallbladder disease
11. Significant pulmonary disorders including: chronic obstructive pulmonary disease, interstitial lung disease, cystic fibrosis, or uncontrolled asthma
12. Regular use of prescription or over-the-counter medications that may affect weight, appetite, food intake, or energy metabolism (e.g. appetite suppressants, lithium, stimulants, anti-psychotics, tricyclic antidepressants; Study M.D. will be consulted as needed; antibiotics started during the intervention period are not an exclusion); regular use of obesity pharmacotherapeutic agents within the last 6 month
13. History of clinically diagnosed eating disorder including anorexia nervosa, bulimia, binge eating disorder
14. Weight loss >5% in past 3 months for any reason except post-partum weight loss; weight gain >5% in past 3 months requires assessment by PI to determine reason for weight gain and if it is appropriate for the subject to participate in the study.
15. Untreated hyper- or hyperthyroidism (TSH outside of normal range for laboratory or history of uncontrolled thyroid disorder). History of thyroid disorder or current thyroid disease treated with stable medication regimen for at least 6 months in acceptable.
16. Current severe depression or history of severe depression within the previous year, based on DSM-IV-TR criteria for Major Depressive Episode.
17. History of other significant psychiatric illness (e.g. psychosis, schizophrenia, mania, bipolar disorder) which in the opinion of the Study MD would interfere with ability to adhere to dietary interventions.
18. Inability to cooperate with/clinical contraindication for MRI including severe claustrophobia, implants, devices, or non-removable body piercings

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2018-06-04 (Actual); Primary Completion 2020-10-13 (Actual); Study Completion 2020-10-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristen Nowak, Ph.D., MPH, Principal Investigator — University of Colorado, Denver
Locations (1):
- Kristen Nowak, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in ADPKD. Data shared will be coded, with no PHI included. Approval of the request and execution of all applicable agreements (i.e. data use agreement) are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol, ICF
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA).

REFERENCES:
- [Derived] St Pierre K, Cashmore BA, Bolignano D, Zoccali C, Ruospo M, Craig JC, Strippoli GF, Mallett AJ, Green SC, Tunnicliffe DJ. Interventions for preventing the progression of autosomal dominant polycystic kidney disease. Cochrane Database Syst Rev. 2024 Oct 2;10(10):CD010294. doi: 10.1002/14651858.CD010294.pub3. PMID 39356039

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant dropped out prior to randomization. This individual is included in the protocol enrollment number, but not the number of participants started.
Period: Overall Study
Arm/Group | Daily Caloric Restriction | Intermittent Fasting
Started | 15 | 13
Completed | 13 | 11
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Daily Caloric Restriction | Intermittent Fasting | Total
Number analyzed (Participants) | 15 | 13 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (12) | 46 (6) | 46 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 16
  Male | 6 | 6 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 14 | 13 | 27
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 14 | 12 | 26
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 13 | 28
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 34.6 (5.1) | 34.8 (5.1) | 34.7 (5.0)
CKD-EPI eGFR [Mean (Standard Deviation); unit: ml/minute/1.73m^2] — Estimated glomerular filtration rate by the Chronic Kidney Disease Epidemiology Collaboration equation. This estimates kidney function. scores of about 90 are normal, where as scores below 60 may indicate kidney disease.
  ml/minute/1.73m^2 | 64 (26) | 75 (16) | 69 (22)
Total Kidney Volume by Magnetic Resonance Imaging (MRI) [Median (Inter-Quartile Range); unit: ml/m] — Height adjusted total kidney volume at baseline by MRI in each group. Population: This baseline measure could not be collected for all participants.
  ml/m
    number analyzed (Participants) | 13 | 12 | 25
    (all) | 994 [589 to 1180] | 835 [476 to 1363] | 916 [476 to 1363]

OUTCOME MEASURES:

1. Primary Outcome: Feasibility to Enroll and Retain Participants
Description: Numbers of individuals pre-screened
Time Frame: Through study completion, an expected duration of 18 months
Measure: Count of Participants; unit: Participants
Groups:
- Overall Study: Pre-screened includes participants that were not randomized.
Arm/Group | Overall Study
Number analyzed (Participants) | 122
Participants | 122

2. Primary Outcome: Feasibility to Enroll Participants
Description: Numbers of individuals screened
Time Frame: Through study completion, an expected duration of 18 months
Measure: Count of Participants; unit: Participants
Groups:
- Overall Study (Screened): Includes all participants screened, whether or not eventually enrolled into either study arm.
Arm/Group | Overall Study (Screened)
Number analyzed (Participants) | 29
Participants | 29

3. Primary Outcome: Feasibility to Retain Participants
Description: Numbers of individuals enrolled
Time Frame: Through study completion, an expected duration of 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Daily Caloric Restriction | Intermittent Fasting
Number analyzed (Participants) | 15 | 13
Participants | 15 | 13

4. Primary Outcome: Feasibility to Retain Participants
Description: Numbers of individuals retained
Time Frame: Through study completion, an expected duration of 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Daily Caloric Restriction | Intermittent Fasting
Number analyzed (Participants) | 15 | 13
Participants | 13 | 11

5. Primary Outcome: Percent Change From Baseline Body Weight (Weight Loss)
Description: Measurement of body weight pre to post intervention in each group
Time Frame: Baseline, 12 weeks, and 1 year
Population: This outcome measure could not be collected for some participants.
Measure: Mean (Standard Deviation); unit: Percent change in weight
Arm/Group | Daily Caloric Restriction | Intermittent Fasting
Number analyzed (Participants) | 12 | 11
Percent change in weight
  12 Weeks | -7.1 (4.2) | -5.5 (3.3)
  1 Year: number analyzed (Participants) | 11 | 11
  1 Year | -9.1 (6.0) | -4.9 (5.6)

6. Secondary Outcome: Safety and Tolerability, Measured as Adverse Events
Description: Number of participants with treatment-related adverse events in each group as evaluated by monthly phone questionnaire
Time Frame: 1 year
Measure: Number; unit: Number of participants w/ adverse events
Arm/Group | Daily Caloric Restriction | Intermittent Fasting
Number analyzed (Participants) | 15 | 13
Number of participants w/ adverse events | 10 | 13

7. Secondary Outcome: Quality of Life Scores at Baseline
Description: Quality of life (QOL) will be assessed with the RAND 36 Item Health Survey (RAND-36) physical and mental health component summary score. The Rand-36 measures quality of life. Possible scores for each subscale range from 0 to 100, with higher scores indicating a better quality of life and better outcome.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Daily Caloric Restriction | Intermittent Fasting
Number analyzed (Participants) | 15 | 13
score on a scale
  Physical Health | 77 (22) | 83 (12)
  Mental Health | 82 (10) | 78 (16)

8. Secondary Outcome: Quality of Life Scores at 12 Weeks
Description: as for outcome 7
Time Frame: 12 Weeks
Population: This outcome measure could not be collected for some participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Daily Caloric Restriction | Intermittent Fasting
Number analyzed (Participants) | 13 | 10
score on a scale
  Physical Health | 81 (21) | 84 (12)
  Mental Health | 80 (26) | 91 (9)

9. Secondary Outcome: Quality of Life Scores at 1 Year
Description: as for outcome 7
Time Frame: 1 Year
Population: This outcome measure could not be collected for some participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Daily Caloric Restriction | Intermittent Fasting
Number analyzed (Participants) | 11 | 11
score on a scale
  Physical Health | 80 (26) | 91 (9)
  Mental Health | 81 (12) | 76 (21)

10. Secondary Outcome: Mood at Baseline
Description: Mood state will be assessed with the Profile of Mood States 2 (POMS-2). The POMS-2 measures mood. Possible scores for the Vigor scale range from 0 to 32, with higher scores for indicating a better outcome. Possible scores for the fatigue scale range from 0 to 28 with higher scores indicating a worse outcome.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Daily Caloric Restriction | Intermittent Fasting
Number analyzed (Participants) | 15 | 13
score on a scale
  Vigor | 8.3 (3.2) | 7.6 (3.0)
  Fatigue | 5.2 (5.4) | 6.4 (3.9)

11. Secondary Outcome: Mood at 12 Weeks
Description: Mood state will be assessed with the Profile of Mood States 2 (POMS-2). The POMS-2 measures mood. Possible scores range from 0 to 20 for both the Vigor and Fatigue subscales, with higher scores indicating a worse outcome.
Time Frame: 12 Weeks
Population: This outcome measure could not be collected for some participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Daily Caloric Restriction | Intermittent Fasting
Number analyzed (Participants) | 13 | 10
score on a scale
  Vigor | 7.5 (3.2) | 7.3 (4.5)
  Fatigue | 7.7 (7.5) | 6.5 (5.4)

12. Secondary Outcome: Mood at 1 Year
Description: as for outcome 11
Time Frame: 1 Year
Population: This outcome measure was not collected for some participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Daily Caloric Restriction | Intermittent Fasting
Number analyzed (Participants) | 11 | 11
score on a scale
  Vigor | 8.2 (4.2) | 7.9 (5.6)
  Fatigue | 5.2 (4.7) | 6.7 (4.8)

13. Secondary Outcome: Change in Energy Intake
Description: Self-reported energy intake
Time Frame: Baseline, 12 weeks and 1 year
Population: This outcome is not reported because the data were not collected.
Arm/Group | Daily Caloric Restriction | Intermittent Fasting
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Change in Macronutrient Intake
Description: Self-reported macronutrient intake
Time Frame: Baseline, 12 weeks and 1 year
Population: This outcome is not reported because the data were not collected.
Arm/Group | Daily Caloric Restriction | Intermittent Fasting
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Serum Insulin-like Growth Factor-1 Levels at Baseline
Description: Serum insulin-like growth factor-1 (IGF-1) levels will be evaluated in each group
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Daily Caloric Restriction | Intermittent Fasting
Number analyzed (Participants) | 15 | 13
ng/ml | 104 (27) | 93 (32)

16. Secondary Outcome: Serum Insulin-like Growth Factor-1 Levels at 12 Weeks
Description: Serum insulin-like growth factor-1 (IGF-1) levels will be evaluated in each group
Time Frame: 12 Weeks
Population: This outcome measure could not be collected for some participants.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Daily Caloric Restriction | Intermittent Fasting
Number analyzed (Participants) | 11 | 11
ng/ml | 127 (41) | 96 (32)

17. Secondary Outcome: Serum Insulin-like Growth Factor-1 Levels at 1 Year
Description: Serum insulin-like growth factor-1 (IGF-1) levels will be evaluated in each group
Time Frame: 1 Year
Population: This outcome measure could not be collected for some participants.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Daily Caloric Restriction | Intermittent Fasting
Number analyzed (Participants) | 10 | 10
ng/ml | 103 (25) | 101 (29)

18. Secondary Outcome: Insulin-like Growth Factor Binding Protein-1 Levels at Baseline
Description: Insulin-like growth factor binding protein-1 (IGFBP-1) levels will be evaluated in each group
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: ng/ml
Arm/Group | Daily Caloric Restriction | Intermittent Fasting
Number analyzed (Participants) | 15 | 13
ng/ml | 9.4 [1.8 to 15.7] | 7.5 [5.2 to 11.2]

19. Secondary Outcome: Insulin-like Growth Factor Binding Protein-1 Levels at 12 Weeks
Description: Insulin-like growth factor binding protein-1 (IGFBP-1) levels will be evaluated in each group
Time Frame: 12 Weeks
Population: This outcome measure could not be collected for some participants.
Measure: Median (Inter-Quartile Range); unit: ng/ml
Arm/Group | Daily Caloric Restriction | Intermittent Fasting
Number analyzed (Participants) | 11 | 11
ng/ml | 11.1 [7.4 to 26.0] | 8.7 [3.1 to 18.8]

20. Secondary Outcome: Insulin-like Growth Factor Binding Protein-1 Levels at 1 Year
Description: Insulin-like growth factor binding protein-1 (IGFBP-1) levels will be evaluated in each group
Time Frame: 1 Year
Population: This outcome measure could not be collected for some participants.
Measure: Median (Inter-Quartile Range); unit: ng/ml
Arm/Group | Daily Caloric Restriction | Intermittent Fasting
Number analyzed (Participants) | 10 | 10
ng/ml | 10.0 [5.8 to 19.6] | 7.9 [4.4 to 10.4]

21. Secondary Outcome: Change in PBMC Ratio of pS6K/s6K
Description: Ratio of protein expression of phosphorylated S6K to S6K peripheral blood mononuclear cell protein expression of S6 kinase (S6K) in each group.
Time Frame: Baseline and 1 year
Population: Not all participants could be analyzed for this outcome measure
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Daily Caloric Restriction | Intermittent Fasting
Number analyzed (Participants) | 6 | 9
ratio
  Baseline | 0.89 (0.39) | 1.43 (1.17)
  Change at 1 year | 0.42 (0.89) | -0.27 (0.58)

22. Secondary Outcome: Change in PBMC pAMPK/AMPK Expression
Description: Ratio of peripheral blood mononuclear cell protein expression of phosphorylated AMP-activated kinase (AMPK) to AMPK in each group
Time Frame: Baseline and 1 year
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Daily Caloric Restriction | Intermittent Fasting
Number analyzed (Participants) | 7 | 9
ratio
  Baseline | 0.49 (0.31) | .76 (0.44)
  Change at 1 Year | 0.12 (0.15) | -0.25 (0.42)

23. Secondary Outcome: Percent Change in Total Kidney Volume by Magnetic Resonance Imaging (MRI)
Description: Percent change from baseline in height adjusted total kidney volume by MRI in each group
Time Frame: Baseline and 1 year
Population: Not all participants could be analyzed for this outcome measure
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Daily Caloric Restriction | Intermittent Fasting
Number analyzed (Participants) | 10 | 10
Percent change | 1.54 (3.35) | 1.70 (6.05)

ADVERSE EVENTS:
Time Frame: 1 Year
Arm/Group | Daily Caloric Restriction | Intermittent Fasting
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/13
Other Adverse Events (participants affected / at risk) | 10/15 | 13/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Daily Caloric Restriction (N=15) | Intermittent Fasting (N=13)
Hunger (Gastrointestinal disorders) | 5 (5) | 11 (11)
Gastrointestinal distress (Gastrointestinal disorders) | 4 (4) | 8 (8)
Fatigue (General disorders) | 1 (1) | 8 (8)
Lightheadedness/dizziness (General disorders) | 3 (3) | 5 (5)
Cold Intolerance (General disorders) | 1 (1) | 7 (7)
Change in mood (Psychiatric disorders) | 2 (2) | 4 (4)
Irritability (Psychiatric disorders) | 1 (1) | 6 (6)
Insomnia (Psychiatric disorders) | 2 (2) | 7 (7)
Headache (Nervous system disorders) | 2 (2) | 4 (4)
Impaired concentration and/or cognitive difficulties (Psychiatric disorders) | 0 (0) | 3 (3)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-05-20): https://cdn.clinicaltrials.gov/large-docs/42/NCT03342742/Prot_SAP_000.pdf
  • Informed Consent Form (2020-03-16): https://cdn.clinicaltrials.gov/large-docs/42/NCT03342742/ICF_001.pdf